CLINICAL TRIAL: NCT06012877
Title: Evaluation of the "Health Friendly" Program to Reduce Children's Fear of the Healthcare Environment.
Acronym: HFriendly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Collaborators: Universidad Pública de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: UPNA-Health_Friendly
Record Dates: First submitted 2023-08-02; First posted 2023-08-28 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Fear
Keywords: Medical Fear; Children; Health Education; Simulated Healthcare Spaces
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial with an intervention group (IG) and a control group (CG) with pre- and post-measurements
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention, known as the Health-Friendly Programme, took place at the Clinical Skills and Simulation Centre of the Public University of Navarre. The intervention consisted of showing the children different scenarios that simulated various medical contexts, letting them experiment with the material and ask questions.
  The structure and content of the intervention were intended to address two main issues. First, the health contexts with which school-age children may come into contact with; these are a consultation at a health centre and a hospital room. Second, the concerns, in relation to intrapersonal, procedural, environmental and interpersonal aspects, experienced by children when they interact with health care professionals or they are sick.
  As reference material, the intervention is described in detail in the guide about the Health-Friendly Programme (Escalada-Hernández et al., 2021).
  Interventions: Behavioral: Health Friendly Program
- Control group (No Intervention): Participants in this group continued with normal activities at school and at home, just like the intervention group, so that the only difference between the two groups was taking part in the intervention. Once the post-study data had been collected from all participants, the participant in the control group also took part in the intervention, a few days later.

INTERVENTIONS:
Behavioral: Health Friendly Program — The intervention, known as the Health-Friendly Programme, took place at the Clinical Skills and Simulation Centre of the Public University of Navarre. The intervention consisted of showing the children different scenarios that simulated various medical contexts, letting them experiment with the material and ask questions.
  The structure and content of the intervention were intended to address two main issues. First, the health contexts with which school-age children may come into contact with; these are a consultation at a health centre and a hospital room. Second, the concerns, in relation to intrapersonal, procedural, environmental and interpersonal aspects, experienced by children when they interact with health care professionals or they are sick.
  As reference material, the intervention is described in detail in the guide about the Health-Friendly Programme (Escalada-Hernández et al., 2021).
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of a novel intervention that involved contact interaction with a simulated healthcare space to reduce medical fear in children in infant class. The main question it aims to answer is: • Will the Health Friendly Program, based on the interaction with a simulate healthcare space, reduce medica fear among children in infant class? Participants will participate in the Health Friendly Program that will consist of showing the children different scenarios that simulated various medical contexts, letting them experiment with the material and ask questions. Researchers will compare two groups (intervention group and control group) to see if there exist differences between both groups in their responses to the Child Medical Fear Scale.

DETAILED DESCRIPTION:
Purpose: This study aimed to evaluate the effectiveness of a novel intervention that involved contact interaction with a simulated healthcare space to reduce medical fear among children in infant class.

Methods: This was an experimental study involving 86 children divided into an intervention group and a control group with pre and post measurements. The intervention, known as the Health-Friendly Programme, consisted of showing children various scenarios that simulated different medical contexts so that they were able to get involved in them, experiment with the materials and ask questions. Medical fear was evaluated using the Spanish version of the revised version of the "Child Medical Fear Scale", which scored fear between 0 and 34 points. The pre-test and post-test levels of medical fear in the intervention and control groups were compared with the Student's t test.

ELIGIBILITY:
Inclusion Criteria:

* Boys and Girls from the third year of Preschool Education (6 years old) at two schools from a town in the North of Spain (school A and B) enrolled in the study.

Exclusion Criteria:

* N/A

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Medical fear | From the participation in the intervention to one week later.
  Medical fear was measured using the revised version of the "Child Medical Fear Scale" (CMFS-R), in its validated Spanish version. The scale has 17 items with statements on fear of certain aspects related to the healthcare environment, that the children answer according to a three-point scale (0 = no fear, 1 = some fear and 2 = very frightened). The maximum total score on the scale is 34 points. The Spanish validation confirmed the existence of the 4 dimensions identified in the original CMFS-R scale: intrapersonal, procedural, environmental and interpersonal fears

CONTACTS AND LOCATIONS:
Overall Officials: Leticia Martín-Rodríguez, PhD, Principal Investigator — Universidad Pública de Navarra
Locations (1):
- Public University of Navarre, Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] San Martin-Rodriguez L, Soto-Ruiz N, Ferraz-Torres M, Garcia-Vivar C, Saralegui-Gainza A, Escalada-Hernandez P. The Spanish Version of the Child Medical Fear Questionnaire: Cross-Cultural Adaptation and Validation. Int J Environ Res Public Health. 2021 Dec 31;19(1):451. doi: 10.3390/ijerph19010451. PMID 35010711